CLINICAL TRIAL: NCT05564377
Title: Molecular Analysis for Combination Therapy Choice (ComboMATCH)
Brief Title: Targeted Therapy Directed by Genetic Testing in Treating Patients With Locally Advanced or Advanced Solid Tumors, The ComboMATCH Screening Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: NCI-2022-06842; NCI-2022-06842 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY191 (Other: ECOG-ACRIN Cancer Research Group); EAY191 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2022-09-27; First posted 2022-10-03 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Advanced Malignant Solid Neoplasm; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Locally Advanced Malignant Solid Neoplasm; Malignant Female Reproductive System Neoplasm; Metastatic HER2-Negative Breast Carcinoma; Metastatic Malignant Solid Neoplasm; Recurrent Endometrial Carcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Malignant Female Reproductive System Neoplasm; Recurrent Malignant Solid Neoplasm; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma; Unresectable HER2-Negative Breast Carcinoma; Unresectable Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis; Endometrial Neoplasms; Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Alpelisib; binimetinib; Biopsy; Specimen Handling; Fluorouracil; dehydroftorafur; Fulvestrant; ipatasertib; Leucovorin; Magnetic Resonance Spectroscopy; neratinib; nilotinib; olaparib; Oxaliplatin; Paclitaxel; Taxes; palbociclib; Panitumumab; sotorasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (20):
- EAY191-A2 (Cohort 1, Arm A) (Experimental): Cohort 1, Arm A: Patients receive olaparib PO BID and alpelisib PO daily on days 1-28 of each cycle. Cycles repeat every 28 days for up to 5 years in the absence of disease progression, unacceptable toxicity, or bone marrow findings consistent with MDS or AML. Patients also undergo MRI, CT, and/or PET scans throughout the trial and a biopsy prior to treatment start. Patients may also undergo bone scans on study as clinically indicated. Patients have the option to also undergo blood collection throughout the trial and a second biopsy at time of disease progression.
  Interventions: Drug: Alpelisib; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Olaparib; Procedure: Positron Emission Tomography
- EAY191-A2 (Cohort 2, Arm B) (Experimental): Cohort 2, Arm B: Patients receive olaparib PO BID and alpelisib PO daily on days 1-28 of each cycle. Cycles repeat every 28 days for up to 5 years in the absence of disease progression, unacceptable toxicity, or bone marrow findings consistent with MDS or AML. Patients also undergo MRI, CT, and/or PET scans throughout the trial and a biopsy prior to treatment start. Patients may also undergo bone scans on study as clinically indicated. Patients have the option to also undergo blood collection throughout the trial and a second biopsy at time of disease progression.
  Interventions: Drug: Alpelisib; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Olaparib; Procedure: Positron Emission Tomography
- EAY191-A2 (Cohort 2, Arm C) (Experimental): Cohort 2, Arm C: Patients receive olaparib PO BID on days 1-28 of each cycle. Cycles repeat every 28 days for up to 5 years in the absence of disease progression, unacceptable toxicity, or bone marrow findings consistent with MDS or AML. Patients experiencing disease progression have the option to migrate to Cohort 3, Arm D. Patients also undergo MRI, CT, and/or PET scans throughout the trial and a biopsy prior to treatment start. Patients may also undergo bone scans on study as clinically indicated. Patients have the option to also undergo blood collection throughout the trial and a second biopsy at time of disease progression.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Olaparib; Procedure: Positron Emission Tomography
- EAY191-A2 (Cohort 3, Arm D) (Experimental): Cohort 3, Arm D: Patients receive olaparib PO BID and alpelisib PO daily on days 1-28 of each cycle. Cycles repeat every 28 days for up to 5 years in the absence of disease progression, unacceptable toxicity, or bone marrow findings consistent with MDS or AML. Patients also undergo MRI, CT, and/or PET scans throughout the trial and a biopsy prior to treatment start. Patients may also undergo bone scans on study as clinically indicated. Patients have the option to also undergo blood collection throughout the trial and a second biopsy at time of disease progression.
  Interventions: Drug: Alpelisib; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Olaparib; Procedure: Positron Emission Tomography
- EAY191-A3 Combo Cohorts 1, 2, 3, 4 (palbociclib, binimetinib) (Experimental): Patients receive palbociclib PO and binimetinib PO throughout the trial. Patients may also undergo biopsy at screening and undergo MRI, CT, bone scan, and collection of blood samples during screening, on study, and/or during follow up.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Palbociclib
- EAY191-A3 Monotherapy Cohort 1 (binimetinib) (Experimental): Patients receive binimetinib PO throughout the trial. Patients may also undergo biopsy at screening and undergo MRI, CT, bone scan, and collection of blood samples during screening, on study, and/or during follow up.
  Interventions: Drug: Binimetinib; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging
- EAY191-A6 Arm I (RAS/RAF/MEK/ERK mutations) (Experimental): Patients receive leucovorin IV, oxaliplatin IV, and fluorouracil IV on study. Patients undergo ECHO and MUGA during screening and on study, a CT with contrast, MRI, or a FDG-PET during screening, collection of blood during screening and on study, and a biopsy during screening. Patients may also undergo brain MRI or CT during screening and on study, bone scans on study, and biopsy on study if clinically indicated.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Echocardiography Test; Drug: Fluorouracil; Drug: Leucovorin; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Drug: Oxaliplatin; Procedure: Positron Emission Tomography
- EAY191-A6 Arm II (RAS/RAF/MEK/ERK mutations) (Experimental): Patients receive binimetinib PO, leucovorin IV, oxaliplatin IV, and fluorouracil IV on study. Patients undergo ECHO and MUGA during screening and on study, a CT with contrast, MRI, or an FDG-PET during screening, collection of blood during screening and on study, and a biopsy during screening. Patients may also undergo brain MRI or CT during screening and on study, bone scans on study, and biopsy on study if clinically indicated
  Interventions: Drug: Binimetinib; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Echocardiography Test; Drug: Fluorouracil; Drug: Leucovorin; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Drug: Oxaliplatin; Procedure: Positron Emission Tomography
- EAY191-E4 (taxane therapy) (Experimental): Patients receive nilotinib hydrochloride monohydrate PO BID on days 1-28 and paclitaxel IV over 1 hour on days 1, 8, and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT or MRI during screening or cycle 1 day 1, every 2 cycles for 1 year, every 3 cycles for patients on study for more than 1 year, and every 4 cycles for patients on study for more than 3 years and may also undergo CT or MRI during follow-up every 3 months for 2 years and then every 6 months for 1 year if clinically indicated. Patients also undergo collection of blood samples at baseline, cycle 2 day 1, and optionally at progression as well as tumor biopsy at baseline and optionally at progression.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Nilotinib Hydrochloride Monohydrate; Drug: Paclitaxel
- EAY191-E5 Cohort I Arm A (sotorasib, panitumumab) (Experimental): Patients receive sotorasib PO QD on days 1-28 and panitumumab IV on days 1 and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood samples, biopsy, and CT or MRI on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Biological: Panitumumab; Drug: Sotorasib
- EAY191-E5 Cohort I Arm B (sotorasib) (Active Comparator): Patients receive sotorasib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression may cross-over to cohort II. Patients also undergo collection of blood samples, biopsy, and CT or MRI on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Sotorasib
- EAY191-E5 Cohort II (sotorasib) (Experimental): Patients receive combination therapy as in EAY191-E5 Arm A.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Biological: Panitumumab; Drug: Sotorasib
- EAY191-N2 Cohort I (Arm I) (NF1 mutations) (Experimental): Patients receive fulvestrant IM on day 1 and day 15 of cycle 1 and day 1 of subsequent cycles and binimetinib PO BID on days 15 to 28 of cycle 1 and day 1 through 28 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo a CT, MRI, or bone scan, ECHO or MUGA, and tumor biopsy, as well as possible blood sample collection during screening and on study.
  Interventions: Drug: Binimetinib; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Echocardiography Test; Drug: Fulvestrant; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan
- EAY191-N2 Cohort I (Arm II) (NF1 mutations) (Experimental): Patients receive fulvestrant IM on day 1 and day 15 of cycle 1 and day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who progress on fulvestrant alone may migrate to cohort II if they meet the migration eligibility criteria. Patients not willing to migrate to cohort II will have further therapy at the investigator's discretion. Patients undergo a CT, MRI, or bone scan and tumor biopsy, as well as ECHO or MUGA and possible blood sample collection during screening and on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Echocardiography Test; Drug: Fulvestrant; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan
- EAY191-N2 Cohort II (NF1 mutations) (Experimental): Patients receive fulvestrant IM on day 1 of each cycle and binimetinib PO BID on days 15-28 of cycle 1 and day 1 through 28 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo a CT, MRI, or bone scan, ECHO or MUGA and tumor biopsy, as well as possible blood sample collection during screening and on study.
  Interventions: Drug: Binimetinib; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Echocardiography Test; Drug: Fulvestrant; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan
- EAY191-N4 Arm I (RAS pathway mutations) (Experimental): Patients receive selumetinib PO BID and olaparib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo a tumor biopsy and blood collection during screening and on study, as well as ECHO or MUGA, and CT scans throughout the trial. Patients may undergo bone marrow aspiration or biopsy as clinically indicated.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Procedure: Mutation Carrier Screening; Drug: Olaparib; Drug: Selumetinib Sulfate
- EAY191-N4 Arm II (RAS pathway mutations) (Active Comparator): Patients receive selumetinib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who experience progression may elect to cross over to Arm I provided they have not had dose limiting toxicities to monotherapy selumetinib. Patients also undergo a tumor biopsy and blood collection during screening and on study, as well as ECHO or MUGA, and CT scans throughout the trial. Patients may undergo bone marrow aspiration or biopsy as clinically indicated.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Procedure: Mutation Carrier Screening; Drug: Selumetinib Sulfate
- EAY191-N5 Arm I (neratinib maleate) (Active Comparator): Patients receive neratinib maleate PO QD on days 1-14 of cycle 0 in the absence of disease progression or unacceptable toxicity. Patients then receive neratinib maleate PO QD on days 1-28 of each subsequent cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who experience progression may crossover to Arm II. Patients undergo ECHO or MUGA during screening and on study, and CT or MRI and collection of blood samples throughout the trial. Patients may also undergo tumor biopsy during screening and on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Drug: Neratinib Maleate
- EAY191-N5 Arm II (neratinib maleate,palbociclib) (Experimental): Patients receive neratinib maleate PO QD on days 1-14 of cycle 0 in the absence of disease progression or unacceptable toxicity. Patients then receive neratinib maleate PO QD on days 1-28 and palbociclib PO QD on days 1-21 of each subsequent cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO or MUGA during screening and on study, and CT or MRI and collection of blood samples throughout the trial. Patients may also undergo tumor biopsy during screening and on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Drug: Neratinib Maleate; Drug: Palbociclib
- EAY191-S3 (activating AKT mutation) (Experimental): Patients receive paclitaxel IV on days 1, 8, and 15 and ipatasertib PO on days 1-21 of each cycle. Treatment repeats every 28 days for up to 35 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo a CT or MRI and blood collection throughout the trial. Patients also undergo a tumor biopsy during screening and optionally during follow-up.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Ipatasertib; Procedure: Magnetic Resonance Imaging; Drug: Paclitaxel

INTERVENTIONS:
Drug: Alpelisib — Given PO
  Other Names: BYL 719; BYL-719; BYL719; Phosphoinositide 3-kinase Inhibitor BYL719; Piqray; VIJOICE
  Arms: EAY191-A2 (Cohort 1, Arm A); EAY191-A2 (Cohort 2, Arm B); EAY191-A2 (Cohort 3, Arm D)
Drug: Binimetinib — Given PO
  Other Names: ARRY 162; ARRY 438162; ARRY-162; ARRY-438162; ARRY162; ARRY438162; MEK 162; MEK-162; MEK162; Mektovi
  Arms: EAY191-A3 Monotherapy Cohort 1 (binimetinib); EAY191-A6 Arm II (RAS/RAF/MEK/ERK mutations); EAY191-N2 Cohort I (Arm I) (NF1 mutations); EAY191-N2 Cohort II (NF1 mutations)
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
  Arms: EAY191-A2 (Cohort 1, Arm A); EAY191-A2 (Cohort 2, Arm B); EAY191-A2 (Cohort 2, Arm C); EAY191-A2 (Cohort 3, Arm D); EAY191-A3 Combo Cohorts 1, 2, 3, 4 (palbociclib, binimetinib); EAY191-A3 Monotherapy Cohort 1 (binimetinib); EAY191-A6 Arm I (RAS/RAF/MEK/ERK mutations); EAY191-E4 (taxane therapy); EAY191-E5 Cohort I Arm A (sotorasib, panitumumab); EAY191-E5 Cohort I Arm B (sotorasib); EAY191-E5 Cohort II (sotorasib); EAY191-N2 Cohort I (Arm I) (NF1 mutations); EAY191-N2 Cohort I (Arm II) (NF1 mutations); EAY191-N2 Cohort II (NF1 mutations); EAY191-N4 Arm I (RAS pathway mutations); EAY191-N4 Arm II (RAS pathway mutations); EAY191-N5 Arm I (neratinib maleate); EAY191-N5 Arm II (neratinib maleate,palbociclib); EAY191-S3 (activating AKT mutation)
Procedure: Biospecimen Collection — Undergo blood collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
  Arms: EAY191-N4 Arm I (RAS pathway mutations); EAY191-N4 Arm II (RAS pathway mutations)
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
  Arms: EAY191-N4 Arm I (RAS pathway mutations); EAY191-N4 Arm II (RAS pathway mutations)
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
  Arms: EAY191-A2 (Cohort 1, Arm A); EAY191-A2 (Cohort 2, Arm B); EAY191-A2 (Cohort 2, Arm C); EAY191-A2 (Cohort 3, Arm D); EAY191-A3 Combo Cohorts 1, 2, 3, 4 (palbociclib, binimetinib); EAY191-A3 Monotherapy Cohort 1 (binimetinib); EAY191-A6 Arm I (RAS/RAF/MEK/ERK mutations); EAY191-A6 Arm II (RAS/RAF/MEK/ERK mutations); EAY191-N2 Cohort I (Arm I) (NF1 mutations); EAY191-N2 Cohort I (Arm II) (NF1 mutations); EAY191-N2 Cohort II (NF1 mutations)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
  Arms: EAY191-A6 Arm I (RAS/RAF/MEK/ERK mutations); EAY191-A6 Arm II (RAS/RAF/MEK/ERK mutations); EAY191-N2 Cohort I (Arm I) (NF1 mutations); EAY191-N2 Cohort I (Arm II) (NF1 mutations); EAY191-N2 Cohort II (NF1 mutations); EAY191-N4 Arm I (RAS pathway mutations); EAY191-N4 Arm II (RAS pathway mutations); EAY191-N5 Arm I (neratinib maleate); EAY191-N5 Arm II (neratinib maleate,palbociclib)
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
  Arms: EAY191-A6 Arm I (RAS/RAF/MEK/ERK mutations); EAY191-A6 Arm II (RAS/RAF/MEK/ERK mutations)
Drug: Fulvestrant — Given IM
  Other Names: Faslodex; Faslodex(ICI 182,780); ICI 182,780; ICI 182780; ICI-182780; ICI182780; ZD 9238; ZD-9238; ZD9238
  Arms: EAY191-N2 Cohort I (Arm I) (NF1 mutations); EAY191-N2 Cohort I (Arm II) (NF1 mutations); EAY191-N2 Cohort II (NF1 mutations)
Drug: Ipatasertib — Given PO
  Other Names: GDC 0068; GDC-0068; GDC0068; RG 7440; RG-7440; RG7440
  Arms: EAY191-S3 (activating AKT mutation)
Drug: Leucovorin — Given IV
  Other Names: Folinic acid
  Arms: EAY191-A6 Arm I (RAS/RAF/MEK/ERK mutations); EAY191-A6 Arm II (RAS/RAF/MEK/ERK mutations)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
  Arms: EAY191-A2 (Cohort 1, Arm A); EAY191-A2 (Cohort 2, Arm B); EAY191-A2 (Cohort 2, Arm C); EAY191-A3 Combo Cohorts 1, 2, 3, 4 (palbociclib, binimetinib); EAY191-A3 Monotherapy Cohort 1 (binimetinib); EAY191-A6 Arm I (RAS/RAF/MEK/ERK mutations); EAY191-A6 Arm II (RAS/RAF/MEK/ERK mutations); EAY191-E4 (taxane therapy); EAY191-E5 Cohort I Arm A (sotorasib, panitumumab); EAY191-E5 Cohort I Arm B (sotorasib); EAY191-E5 Cohort II (sotorasib); EAY191-N2 Cohort I (Arm I) (NF1 mutations); EAY191-N2 Cohort I (Arm II) (NF1 mutations); EAY191-N2 Cohort II (NF1 mutations); EAY191-N5 Arm I (neratinib maleate); EAY191-N5 Arm II (neratinib maleate,palbociclib); EAY191-S3 (activating AKT mutation)
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
  Arms: EAY191-A6 Arm I (RAS/RAF/MEK/ERK mutations); EAY191-A6 Arm II (RAS/RAF/MEK/ERK mutations); EAY191-N2 Cohort I (Arm I) (NF1 mutations); EAY191-N2 Cohort I (Arm II) (NF1 mutations); EAY191-N2 Cohort II (NF1 mutations); EAY191-N4 Arm I (RAS pathway mutations); EAY191-N4 Arm II (RAS pathway mutations); EAY191-N5 Arm I (neratinib maleate); EAY191-N5 Arm II (neratinib maleate,palbociclib)
Procedure: Mutation Carrier Screening — Undergo tumor mutational screening
  Arms: EAY191-N4 Arm I (RAS pathway mutations); EAY191-N4 Arm II (RAS pathway mutations)
Drug: Neratinib Maleate — Given PO
  Other Names: 2-Butenamide, N-(4-((3-chloro-4-(2-pyridinylmethoxy)phenyl)amino)-3-cyano-7-ethoxy-6-quinolinyl)-4-(dimethylamino)-, (2E)-, (2Z)-2-butenedioate (1:1); HKI-272 Maleate; NERATINIB MALEATE ANHYDROUS; Nerlynx
  Arms: EAY191-N5 Arm I (neratinib maleate); EAY191-N5 Arm II (neratinib maleate,palbociclib)
Drug: Nilotinib Hydrochloride Monohydrate — Given PO
  Other Names: AMN 107; AMN-107; AMN107; Nilotinib Monohydrochloride Monohydrate; Tasigna
  Arms: EAY191-E4 (taxane therapy)
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU 0059436; KU-0059436; KU0059436; Lynparza; Olanib; Olaparix; PARP Inhibitor AZD2281
  Arms: EAY191-A2 (Cohort 1, Arm A); EAY191-A2 (Cohort 2, Arm B); EAY191-A2 (Cohort 2, Arm C); EAY191-A2 (Cohort 3, Arm D); EAY191-N4 Arm I (RAS pathway mutations)
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; Elplat; JM 83; JM-83; JM83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; RP54780; SR 96669; SR-96669; SR96669
  Arms: EAY191-A6 Arm I (RAS/RAF/MEK/ERK mutations); EAY191-A6 Arm II (RAS/RAF/MEK/ERK mutations)
Drug: Paclitaxel — Given PO or IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: EAY191-E4 (taxane therapy); EAY191-S3 (activating AKT mutation)
Drug: Palbociclib — Given PO
  Other Names: 6-Acetyl-8-cyclopentyl-5-methyl-2-((5-(piperazin-1-yl)pyridin-2-yl)amino)-8h-pyrido(2,3-d)pyrimidin-7-one; Ibrance; PD 0332991; PD 332991; PD 991; PD-0332991; PD0332991
  Arms: EAY191-A3 Combo Cohorts 1, 2, 3, 4 (palbociclib, binimetinib); EAY191-N5 Arm II (neratinib maleate,palbociclib)
Biological: Panitumumab — Given IV
  Other Names: ABX-EGF; ABX-EGF Monoclonal Antibody; ABX-EGF, Clone E7.6.3; E7.6.3; Human IgG2K Monoclonal Antibody; MoAb ABX-EGF; MoAb E7.6.3; Monoclonal Antibody ABX-EGF; Monoclonal Antibody E7.6.3; Vectibix
  Arms: EAY191-E5 Cohort I Arm A (sotorasib, panitumumab); EAY191-E5 Cohort II (sotorasib)
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
  Arms: EAY191-A2 (Cohort 1, Arm A); EAY191-A2 (Cohort 2, Arm B); EAY191-A2 (Cohort 2, Arm C); EAY191-A2 (Cohort 3, Arm D); EAY191-A6 Arm I (RAS/RAF/MEK/ERK mutations); EAY191-A6 Arm II (RAS/RAF/MEK/ERK mutations)
Drug: Selumetinib Sulfate — Given PO
  Other Names: AZD-6244 Hydrogen Sulfate; AZD6244 Hydrogen Sulfate; AZD6244 Hydrogen Sulphate; Koselugo; Selumetinib Sulphate
  Arms: EAY191-N4 Arm I (RAS pathway mutations); EAY191-N4 Arm II (RAS pathway mutations)
Drug: Sotorasib — Given PO
  Other Names: AMG 510; AMG-510; AMG510; Lumakras; Lumykras
  Arms: EAY191-E5 Cohort I Arm A (sotorasib, panitumumab); EAY191-E5 Cohort I Arm B (sotorasib); EAY191-E5 Cohort II (sotorasib)

SUMMARY:
This ComboMATCH patient screening trial is the gateway to a coordinated set of clinical trials to study cancer treatment directed by genetic testing. Patients with solid tumors that have spread to nearby tissue or lymph nodes (locally advanced) or have spread to other places in the body (advanced) and have progressed on at least one line of standard systemic therapy or have no standard treatment that has been shown to prolong overall survival may be candidates for these trials. Genetic tests look at the unique genetic material (genes) of patients' tumor cells. Patients with some genetic changes or abnormalities (mutations) may benefit from treatment that targets that particular genetic mutation. ComboMATCH is designed to match patients to a treatment that may work to control their tumor and may help doctors plan better treatment for patients with locally advanced or advanced solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To register, allocate, and assign patients to ComboMATCH treatment trials.

SECONDARY OBJECTIVES:

I. To evaluate the rate of positive outcomes in defined cohorts within treatment trials of treatment combinations including targeted therapies for molecularly defined populations, and also in the subset of treatment trials where the treatments are supported by in vivo models.

II. To perform quality control of the patients registered in the form of pathological confirmation of disease and sub-type to confirm diagnosis and treatment arm allocation.

SECONDARY CORRELATIVE OBJECTIVES:

I. Assess the concordance of the central molecular characterization of the pre-treatment biopsy samples with the genetic readouts from the Designated Laboratories (DLs) for patients enrolled on the ComboMATCH treatment trials.

II. To assess how the registration diagnostic tumor mutation profile and pre-treatment biopsy profile compare to the circulating tumor-derived deoxyribonucleic acid (ctDNA) mutation profile from plasma.

EXPLORATORY OBJECTIVE:

I. Assess association between ComboMATCH treatment trials outcomes (positive or negative) with the type of rationale for the selected drug combinations and the type of rationale for the gene variant/combination for selection (e.g., whether the trial was based on targeted therapies for molecularly defined populations, those that were supported by in vivo models, and those that were supported by empiric clinical data).

OUTLINE:

REGISTRATION: Patients undergo tumor mutational screening of previously-collected tumor samples for specific, pre-defined mutations, amplifications, or translocations of interest via tumor sequencing. Patients who are 18 years or older and have biopsiable disease undergo a new biopsy for research purposes prior to initiating treatment on the ComboMATCH treatment trial.

TREATMENT: Patients with mutations targeted to investigational combination therapies are assigned to 1 of 20 treatment subprotocols.

EAY191-N4: Patients with RAS pathway mutant ovarian or endometrial cancer are randomized to 1 of 2 arms.

ARM I: Patients receive selumetinib orally (PO) twice daily (BID) and olaparib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo a tumor biopsy and blood collection during screening and on study, as well as echocardiogram (ECHO) or multigated acquisition (MUGA), and computed tomography (CT) scans throughout the trial. Patients may undergo bone marrow aspiration or biopsy as clinically indicated.

ARM II: Patients receive selumetinib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who experience progression may elect to cross over to Arm I provided they have not had dose limiting toxicities to monotherapy selumetinib. Patients also undergo a tumor biopsy and blood collection during screening and on study, as well as ECHO or MUGA, and CT scans throughout the trial. Patients may undergo bone marrow aspiration or biopsy as clinically indicated.

EAY191-N2: Patients with inactivating or inferred inactivating NF1 alterations, and hormone receptor positive, HER2-negative metastatic breast cancer. Patients who are fulvestrant naive are assigned to Cohort I, while patients who are fulvestrant resistant are assigned to Cohort II.

COHORT I: Patients are randomized to 1 of 2 arms.

ARM I:Patients receive fulvestrant intramuscularly (IM) on day 1 and day 15 of cycle 1 and day 1 of subsequent cycles and binimetinib PO BID on days 15 to 28 of cycle 1 and day 1 through 28 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo a CT, magnetic resonance imaging (MRI), or bone scan, ECHO or MUGA, and tumor biopsy, as well as possible blood sample collection during screening and on study.

ARM II: Patients receive fulvestrant IM on day 1 and day 15 of cycle 1 and day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who progress on fulvestrant alone may migrate to cohort II if they meet the migration eligibility criteria. Patients not willing to migrate to cohort II will have further therapy at the investigator's discretion. Patients undergo a CT, MRI, or bone scan and tumor biopsy, as well as ECHO or MUGA and possible blood sample collection during screening and on study.

COHORT II: Patients receive fulvestrant IM on day 1 of each cycle and binimetinib PO BID on days 15-28 of cycle 1 and day 1 through 28 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo a CT, MRI, or bone scan, ECHO or MUGA and tumor biopsy, as well as possible blood sample collection during screening and on study.

EAY191-E4: Patients with solid tumors who previously underwent taxane therapy.

Patients receive nilotinib hydrochloride monohydrate PO BID on days 1-28 and paclitaxel intravenously (IV) over 1 hour on days 1, 8, and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT or MRI during screening or cycle 1 day 1, every 2 cycles for 1 year, every 3 cycles for patients on study for more than 1 year, and every 4 cycles for patients on study for more than 3 years and may also undergo CT or MRI during follow-up every 3 months for 2 years and then every 6 months for 1 year if clinically indicated. Patients also undergo collection of blood samples at baseline, cycle 2 day 1, and optionally at progression as well as tumor biopsy at baseline and optionally at progression.

EAY191-A3: Patients with KRAS/NRAS/BRAF mutated low-grade serous ovarian cancer (LGSOC) naive to MEK or CDK4/6 inhibitor therapy are randomized to either combination cohort 1 or monotherapy cohort 1. Patients with LGSOC who have received prior MEK inhibitor therapy are assigned to combination cohort 2. Patients with KRAS/NRAS/HRAS/non-V600E BRAF mutated pancreatic cancer are assigned to combination cohort 3. Patients with all other KRAS/NRAS/HRAS mutated tumor types (excluding LGSOC, non-small cell lung cancer, colorectal cancer, pancreatic, and melanoma) are assigned to combination cohort 4.

COMBINATION COHORTS 1, 2, 3, 4: Patients receive palbociclib PO and binimetinib PO throughout the trial. Patients may also undergo biopsy at screening and undergo MRI, CT, bone scan, and collection of blood samples during screening, on study, and/or during follow up.

MONOTHERAPY COHORT 1: Patients receive binimetinib PO throughout the trial. Patients may also undergo biopsy at screening and undergo MRI, CT, bone scan, and collection of blood samples during screening, on study, and/or during follow up.

EAY191-S3: Patients with an activating AKT mutation solid tumor.

Patients receive paclitaxel IV on days 1, 8, and 15 and ipatasertib PO on days 1-21 of each cycle. Treatment repeats every 28 days for up to 35 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo a CT or MRI and blood collection throughout the trial. Patients also undergo a tumor biopsy during screening and optionally during follow-up.

EAY191-A6: Patients with RAS/RAF/MEK/ERK mutant biliary tract cancers are randomized to 1 of 2 arms.

ARM 1: Patients receive leucovorin IV, oxaliplatin IV, and fluorouracil IV on study. Patients undergo echocardiogram (ECHO) and multigated acquisition scan (MUGA) during screening and on study, a CT with contrast, MRI, or a fludeoxyglucose F-18 positron emission tomography (FDG-PET) during screening, collection of blood during screening and on study, and a biopsy during screening. Patients may also undergo brain MRI or CT during screening and on study, bone scans on study, and biopsy on study if clinically indicated.

ARM 2: Patients receive binimetinib PO, leucovorin IV, oxaliplatin IV, and fluorouracil IV on study. Patients undergo ECHO and MUGA during screening and on study, a CT with contrast, MRI, or an FDG-PET during screening, collection of blood during screening and on study, and a biopsy during screening. Patients may also undergo brain MRI or CT during screening and on study, bone scans on study, and biopsy on study if clinically indicated.

EAY191-E5: Patients are assigned to 1 of 2 cohorts.

COHORT I: Patients who have never received a KRAS G12C inhibitor are randomized to arms A or B.

ARM A: Patients receive sotorasib PO once daily (QD) on days 1-28 and panitumumab intravenously IV on days 1 and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood samples, biopsy, and CT or MRI on study.

ARM B: Patients receive sotorasib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression may cross-over to cohort II. Patients also undergo collection of blood samples, biopsy, and CT or MRI on study.

COHORT II: Patients who have received a KRAS G12C inhibitor are assigned to arm C.

ARM C: Patients receive combination therapy as in Arm A.

EAY191-A2: Patients are assigned to 1 of 3 cohorts.

COHORT 1: PARP-inhibitor naive patients are assigned to Arm A.

ARM A: Patients receive olaparib PO BID and alpelisib PO daily on days 1-28 of each cycle. Cycles repeat every 28 days for up to 5 years in the absence of disease progression, unacceptable toxicity, or bone marrow findings consistent with myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML). Patients also undergo MRI, CT, and/or PET scans throughout the trial and a biopsy prior to treatment start. Patients may also undergo bone scans on study as clinically indicated. Patients have the option to also undergo blood collection throughout the trial and a second biopsy at time of disease progression.

COHORT 2: PARP-inhibitor naive patients are randomized to 1 of 2 arms.

ARM B: Patients receive olaparib PO BID and alpelisib PO daily on days 1-28 of each cycle. Cycles repeat every 28 days for up to 5 years in the absence of disease progression, unacceptable toxicity, or bone marrow findings consistent with MDS or AML. Patients also undergo MRI, CT, and/or PET scans throughout the trial and a biopsy prior to treatment start. Patients may also undergo bone scans on study as clinically indicated. Patients have the option to also undergo blood collection throughout the trial and a second biopsy at time of disease progression.

ARM C: Patients receive olaparib PO BID on days 1-28 of each cycle. Cycles repeat every 28 days for up to 5 years in the absence of disease progression, unacceptable toxicity, or bone marrow findings consistent with MDS or AML. Patients experiencing disease progression have the option to migrate to Cohort 3, Arm D. Patients also undergo MRI, CT, and/or PET scans throughout the trial and a biopsy prior to treatment start. Patients may also undergo bone scans on study as clinically indicated. Patients have the option to also undergo blood collection throughout the trial and a second biopsy at time of disease progression.

COHORT 3: PARP-inhibitor resistant patients are assigned to Arm D.

ARM D: Patients receive olaparib PO BID and alpelisib PO daily on days 1-28 of each cycle. Cycles repeat every 28 days for up to 5 years in the absence of disease progression, unacceptable toxicity, or bone marrow findings consistent with MDS or AML. Patients also undergo MRI, CT, and/or PET scans throughout the trial and a biopsy prior to treatment start. Patients may also undergo bone scans on study as clinically indicated. Patients have the option to also undergo blood collection throughout the trial and a second biopsy at time of disease progression.

EAY191-N5: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive neratinib maleate PO QD on days 1-14 of cycle 0 in the absence of disease progression or unacceptable toxicity. Patients then receive neratinib maleate PO QD on days 1-28 of each subsequent cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who experience progression may crossover to Arm II. Patients undergo ECHO or MUGA during screening and on study, and CT or MRI and collection of blood samples throughout the trial. Patients may also undergo tumor biopsy during screening and on study.

ARM II: Patients receive neratinib maleate PO QD on days 1-14 of cycle 0 in the absence of disease progression or unacceptable toxicity. Patients then receive neratinib maleate PO QD on days 1-28 and palbociclib PO QD on days 1-21 of each subsequent cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO or MUGA during screening and on study, and CT or MRI and collection of blood samples throughout the trial. Patients may also undergo tumor biopsy during screening and on study.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have measurable disease
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status between 0-2 OR patient must have Lansky performance status of >= 50% or Karnofsky performance status of >= 50%
* Patient must be deemed potentially eligible for a ComboMATCH Treatment Trial as assessed by the enrolling provider
* All patients must have sequencing results available from a National Cancer Institute (NCI) credentialed Designated Laboratory (DL)
* Patients must have locally advanced or advanced histologically documented solid tumors requiring therapy and meet one of the following criteria:

  * Patients must have progressed on at least one line of standard systemic therapy OR
  * Patients whose disease has no standard treatment that has been shown to prolong overall survival
* Patient must meet one of the following requirements:

  * Patients 18 years and older who have tumor amenable to minimal risk image-guided or direct vision biopsy and must be willing and able to undergo a tumor biopsy to obtain samples for research if the patient is to enroll in a ComboMATCH treatment trial OR
  * Patients 18 years and older who do not have disease that is biopsiable at minimal risk to the patient must confirm availability of an archival tumor tissue specimen for submission for research if the patient enrolls to a ComboMATCH Treatment Trial. This tumor tissue must meet the following criteria:

    * Tissue must have been collected within 12 months prior to registration to the EAY191 Registration Trial
    * Patient must not have had a Response Evaluation Criteria in Solid Tumors (RECIST) response (complete response [CR] or partial response [PR]) to any intervening therapy after collection of the tissue
    * Formalin-fixed paraffin-embedded tumor tissue block(s) or slides must be available OR
  * Patients under 18 years old must confirm availability of an archival tumor tissue specimen for submission for research if patient enrolls to a ComboMATCH Treatment Trial. This tumor tissue must meet the following criteria:

    * Formalin-fixed paraffin-embedded tumor tissue block(s) or slides must be available
  * NOTE: See specific ComboMATCH Treatment Trial protocol for tissue collection and management instructions. Performance of the mandatory research biopsy or submission of pre-trial formalin-fixed paraffin-embedded (FFPE) and collection and submission of the blood specimens for the integrated studies will be performed under the consent authority of the specific treatment trial protocol to which the patient is registered. No procedures to collect specimens for research only are to be performed for patients registered to the EAY191 Registration Trial only
* NOTE: Each ComboMATCH Treatment Trial contains specific eligibility criteria. If patient is found to not be eligible for the assigned ComboMATCH Treatment Trial, indication of ineligibility will trigger re-evaluation and potential assignment to another Treatment Trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2900 (Estimated)
Dates: Start 2023-04-07 (Actual); Primary Completion 2030-07-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
Accrual of patients to ComboMATCH treatment trials | Up to 8 years
  Will be estimated over time and considered in relationship to changes in treatment trial cohort status (activations, suspensions, terminations).
Assignment of patients to ComboMATCH treatment trials | Up to 8 years
  Will be estimated over time and considered in relationship to changes in treatment trial cohort status (activations, suspensions, terminations).
Enrollment rates to ComboMATCH treatment trials | Up to 8 years
  Will be estimated over time and considered in relationship to changes in treatment trial cohort status (activations, suspensions, terminations).

SECONDARY OUTCOMES:
Rate of positive outcomes within the treatment trial defined cohorts | Up to 8 years
  For each cohort in each treatment trial there is a defined primary efficacy endpoint (usually progression free survival [PFS] or overall response rate) and defined primary analysis for evaluating the primary endpoint. As cohorts are completed, whether they meet the criteria for a positive primary outcome will be determined. Positive treatment cohort outcome (on primary endpoint) will be analyzed as a binary random variable. The raw proportion of treatment cohorts with positive outcomes and an exact binomial confidence interval will be computed. If there are a sufficient number of treatment cohorts, logistic regression analysis will be performed examining the relationship of treatment cohort characteristics with successful outcomes. The goal is to achieve a rate of at least 30% with positive outcomes, both overall and in the subset of treatment trials based on in vivo models.

OTHER OUTCOMES:
Concordance between whole exome sequencing (WES) and results from the Designated Laboratory (DL) | Up to 8 years
  Whole exome and other sequencing will be performed on mandatory tissue biopsies or, if no biopsy tissue is available, on submitted formalin-fixed paraffin-embedded tissue. These assays will be done in a clinical laboratory (e.g., Clinical Laboratory Improvement Act-compliant); but results will not be returned to the clinical site. Results will be used to compare with the DL assay results. This comparison will be required to conduct an important secondary analysis of the primary endpoint in each cohort in each treatment trial, restricting to those cases that are concordant between WES and the result from the DL that was the basis for enrollment (integrated).

CONTACTS AND LOCATIONS:
Overall Officials: James M Ford, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (470):
- United States (466):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - Kingman Regional Medical Center, Kingman, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - PCR Oncology, Arroyo Grande, California
  - Mercy Cancer Center - Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Epic Care-Dublin, Dublin, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - UC San Diego Health System - Encinitas, Encinitas, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - The Angeles Clinic and Research Institute - West Los Angeles Office, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Children's Hospital of Orange County, Orange, California
  - Saint Joseph Hospital - Orange, Orange, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - Sharp Memorial Hospital, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Saint John's Cancer Institute, Santa Monica, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - Presbyterian Intercommunity Hospital, Whittier, California
  - Woodland Memorial Hospital, Woodland, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - CTCA at Southeastern Regional Medical Center, Newnan, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Mercyhealth Cancer Institute - Rockford, Rockford, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Mercy Health - Paducah Cancer Center, Paducah, Kentucky
  - East Jefferson General Hospital, Metairie, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - UPMC Western Maryland, Cumberland, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Tufts Medical Center Cancer Center Stoneham, Stoneham, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - University of Michigan - Brighton Center for Specialty Care, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Gulfport Memorial Hospital, Gulfport, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Hunterdon Medical Center, Flemington, New Jersey
  - Monmouth Medical Center Southern Campus, Lakewood, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Capital Health Medical Center-Hopewell, Pennington, New Jersey
  - Sidney Kimmel Cancer Center Washington Township, Sewell, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Pluta Cancer Center, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Cone Health MedCenter Asheboro, Asheboro, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Cone Health Cancer Center at Drawbridge Parkway, Greensboro, North Carolina
  - Hayworth Cancer Center, High Point, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Duke Women's Cancer Care Raleigh, Raleigh, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - UH Seidman Cancer Center at UH Avon Health Center, Avon, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Columbus Oncology and Hematology Associates, Dublin, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Zangmeister Center Grove City, Grove City, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Memorial Hospital, Marysville, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC Altoona, Altoona, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Roger Williams Medical Center, Providence, Rhode Island
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Hendrick Medical Center, Abilene, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Methodist Willowbrook Hospital, Houston, Texas
  - Houston Methodist West Hospital, Houston, Texas
  - Covenant Medical Center-Lakeside, Lubbock, Texas
  - Houston Methodist Saint John Hospital, Nassau Bay, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - Houston Methodist The Woodlands Hospital, The Woodlands, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Valley Medical Center, Renton, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - ThedaCare Regional Medical Center - Appleton, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - ThedaCare Cancer Care - Berlin, Berlin, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercyhealth Hospital and Cancer Center - Janesville, Janesville, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ThedaCare Regional Medical Center - Neenah, Neenah, Wisconsin
  - ThedaCare Cancer Care - New London, New London, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - ThedaCare Cancer Care - Oshkosh, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - ThedaCare Cancer Care - Shawano, Shawano, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Sheboygan Physicians Group, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - ThedaCare Cancer Care - Waupaca, Waupaca, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
- Puerto Rico (4):
  - Puerto Rico Hematology Oncology Group, Bayamón
  - Doctors Cancer Center, Manatí
  - Centro Comprensivo de Cancer de UPR, San Juan
  - PROncology, San Juan

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm